CLINICAL TRIAL: NCT04970420
Title: Evaluation of Nursing Interventions Given to Immigrant Women (Ahıska Turks) Towards Health Responsibility, Family Planning Knowledge and Attitude
Brief Title: Health Responsibility and Family Planning ın Immigrant Women (Ahıska Turks).
Acronym: HeRFAPIW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ezgi Demirtürk Selçuk, Academician, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0061
Record Dates: First submitted 2021-06-30; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Health, Subjective; Family Planning; Women; Nurse
Keywords: Family planning; Knowledge; Emigration; Attitude; Immigration
MeSH Terms: conditions — Behavior | interventions — Family Planning Services; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeRFAPIW (Experimental): Health Responsibility and Family Planning ın Immigrant Women (Ahıska Turks).
  Interventions: Other: Health Responsibility and Family Planning ın Immigrant Women (Ahıska Turks).
- Control group (Active Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Health Responsibility and Family Planning ın Immigrant Women (Ahıska Turks). — In this study, individual training, training via mobile application and telephone counseling will be given to the experimental group. During the meetings, attention will be paid to the pandemic rules.
  Arms: HeRFAPIW
Other: Control group — Individual training, mobile application and telephone counseling will be given to the control group after the study data is collected.
  Arms: Control group

SUMMARY:
Purpose: The aims of the research are to determine the effects of individual trainings on family planning given to migrant women (Ahıska Turks), repetitive trainings via mobile applications, telephone counseling initiatives on women's health responsibility levels, family planning knowledge and attitudes.

Design: This pretest-posttest is an interventional quasi-experimental research. Method: Standard protocol Items: Recommendations for Interventional Trials (SPIRIT) Statement 2013 checklist is used in this study. The CONSORT (Consolidated Standards of Reporting Trials) flowchart is used in this protocol. This study will be carried out with immigrant (Ahıska Turks) women between the ages of 15-49 who are registered in Üzümlü Family Health Center in Üzümlü district of Erzincan province. In this study, individual training on family planning and health responsibility, repetitive training via mobile application and telephone counseling initiatives will be made. The same applications will be applied to the control group after the study data is collected.

Hypotheses: H1: Mobile applications for family planning, telephone counseling and individual training have an impact on the family planning attitudes of immigrant women.

H1: Mobile applications for family planning, telephone counseling and individual trainings have an impact on the family planning knowledge level of immigrant women.

H1: Mobile applications, telephone counseling and individual trainings for health responsibility have an impact on the level of health responsibility of migrant women.

ELIGIBILITY:
Inclusion Criteria:

* To be registered at the family health center
* Being literate
* Ability to communicate verbally
* Volunteering to participate in the research
* Owning a smartphone or a phone belonging to any member of the family that can also be used by the participant
* Having internet access at home or at work
* Internet use
* Able to speak and write Turkish
* Being a migrant woman in the age group of 15-49

Exclusion Criteria:

* Having a physical or mental health problem
* Menopausal, tubal ligation or spouse vasectomy
* Inability to reach by phone/visit
* Relocation of women to another place
* Illness and death of the sampled woman
* To have received training on effective family planning

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 86 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors Scale II-Health Responsibility Sub-Dimension | Change in health responsibility at baseline and after 12 weeks.
  The lowest score in the Health Responsibility Sub-Dimension was determined as 9 and the highest as 36 points. As the score obtained from the Sub-Dimension of the Scale increases, the health responsibility increases. Health Responsibility sub-dimension Cronbach Alpha coefficient is 0.77.
Family Planning Attitude Scale | Change in health responsibility at baseline and after 12 weeks.
  A minimum of 34 and a maximum of 170 points can be obtained from the scale. The scale has 3 sub-dimensions: "Attitude of the Society towards Family Planning", "Attitude towards Family Planning Methods" and "Attitude towards Birth". Evaluation of the scale is done as individuals with higher scores have more positive family planning attitudes. The internal consistency and homogeneity coefficients determined by the alpha correlations of the scale were found to be 0.90 in total.
Family Planning Information Form | Change in health responsibility at baseline and after 12 weeks.
  This form, which was developed by the researcher based on the literature, consists of questions that include mobile application and telephone counseling comprehensive initiatives. A minimum of 0 and a maximum of 75 points are taken from the form. Evaluation of the form is made as individuals with high scores have knowledge about family planning.

SECONDARY OUTCOMES:
Family Planning Program Evaluation Form | Level of satisfaction with the programs implemented after 12 weeks
  In the form developed by the researchers, it is related to the benefits of the family planning training program for the participants, their satisfaction with the training program, the perception of the knowledge level of women on family planning after the training, suggestions for the development of the training program and the family planning method used after the training. There are 7 questions.

IPD SHARING:
Plan to Share IPD: No